CLINICAL TRIAL: NCT00161018
Title: New Antipsychotic Strategies: Quetiapine and Risperidone vs. Fluphenazine in Treatment Resistant Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, MPRC, PI, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-20725
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Risperidone; Fluphenazine

INTERVENTIONS:
Drug: Quetiapine, Risperidone, Fluphenazine

SUMMARY:
The purpose of this study is to:

1. Evaluate the efficacy and safety of the new antipsychotics, quetiapine (300-500mg/day) and risperidone (3-4mg/day) compared to each other and to fluphenazine (10-15mg/day), a high potency typical antipsychotic in patients who meet the DSM IV criteria for schizophrenia.
2. To evaluate the efficacy and safety of quetiapine (1200mg/day) in patients who have not responded to conventional and newer antipsychotics.
3. To evaluate the effectiveness of quetiapine (300-500mg/day), and risperidone (3-5mg/day) compared to each other and fluphenazine (10-15mg/day) in the treatment of hostility and aggression in treatment-resistant schizophrenic patients.
4. To evaluate the effectiveness of quetiapine (300-500mg/day) and risperidone (3-5mg/day) compared to each other and fluphenazine (10-15mg/day) on rates of discharge, quality of life, and independent living skills.
5. To assess prolactin levels and to evaluate any relationship with sexual dysfunction and menstrual irregularities.
6. To evaluate the possible differential impact of treatment conditions on cognitive functioning including measures of attention, motor speed, problem solving, verbal and visual memory, and verbal processing speed.
7. To measure changes in weight and health consequences associated with weight changes.

DETAILED DESCRIPTION:
This is a three arm multi-center randomized double-blind study. After open label treatment with each individual being optimized with routine antipsychotic treatment for 4-6 weeks to prospectively establish lack of response to conventional antipsychotic therapy, approximately 180 patients with schizophrenia who are experiencing clinically significant psychotic symptoms will be recruited (minimum 150 enrolled) in the double-blind period of the study. All participants will sign consent forms before participating in this research study. If participants choose to enroll in the high dose quetiapine arm (period IIIb), they will sign an additional consent form before entering period IIIb.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, between ages 18 and 65 year sof age.
* Females of childbearing potential must agree to use medically accepted means of contraception.
* A diagnosis of schizophrenia according to the DSM-IV.
* Subjects must meet retrospective criteria for treatment-resistance as defined:

  1. Persistent positive psychotic symptoms.
  2. Current presence of at least a moderately severe illness as rated by the total BPRS.
  3. Persistence of illness- No evidence of good functioning in the last five years.
  4. Drug-refectory condition defined as at least two periods of treatment in the preceding significant symptom relief.
* Subjects must been judged competent to consent by the ESC evaluation and provide voluntary informed consent.
* Subjects must be reliable. They must agree to cooperate with all tests and examinations required by the protocol.
* Patients msut have a normal ophthalmoscopic exam within 6 months of a full eye exam if any lense abnormality prior to entering study.

Exclusion Criteria:

* Females who are either pregnant or lactating.
* Serious medical illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease such that hospitalization for the disease is anticipated within three months or death is anticipated with three years.
* History of severe allergies or multiple adverse drug reactions.
* DSM-IV substance abuse or dependence within the past month.
* Any DSM-IV organic mental disorder.
* Judged clinically to be at serious suicidal risk.
* Definitive failure to show clinically significant response (improved in CGI score of at least 1 point) to and adequate trial of clozapine (600mg/day for at least 6 weeks)
* Uncontrolled seizures within the past 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-11 (Actual); Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of the new antipsychotics, quetiapine(300-500mg/day) and risperidone(3-5mg/day) compared to each other and to fluphenazine(10-15mg/day), a high potency typical antipsychotic

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Conley, MD, Principal Investigator — MPRC
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States